CLINICAL TRIAL: NCT04349930
Title: The CBD-IC Randomized Controlled Trial: Evaluation of Hemp Cannabidiol SuppositoRies for Pain and Urinary SymptOms in INterstitial Cystitis (CHRONIC)
Acronym: CHRONIC
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Need to obtain IND approval.
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Gena Dunivan, M.D, Associate Professor, University of New Mexico
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 00-000
Record Dates: First submitted 2020-04-13; First posted 2020-04-16 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Interstitial Cystitis; Bladder Pain Syndrome
Keywords: Interstitial cystitis; Bladder pain syndrome; IC; BPS; CBD; Cannabidiol; Hemp
MeSH Terms: conditions — Cystitis, Interstitial

STUDY DESIGN:
Intervention Model Description: Double-masked, placebo-controlled randomized trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-masked (patient and provider)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cannabidiol (Experimental): CBD vaginal suppository
  Interventions: Drug: Cannabidiol vaginal suppository
- Placebo (Placebo Comparator): Placebo vaginal suppository
  Interventions: Drug: Placebo vaginal suppository

INTERVENTIONS:
Drug: Cannabidiol vaginal suppository — Cannabidiol vaginal suppository
  Arms: Cannabidiol
Drug: Placebo vaginal suppository — Placebo vaginal suppository
  Arms: Placebo

SUMMARY:
This study seeks to exploit bladder cannabidiol receptors as a therapeutic drug target by conducting a double-masked, placebo-controlled randomized trial evaluating the effects of vaginal hemp cannabidiol (CBD) suppositories on lower urinary tract symptoms (LUTS), pain severity, and sexual function.

DETAILED DESCRIPTION:
Interstitial Cystitis/Bladder Pain Syndrome (IC/BPS) is a chronic inflammatory disease with an insidious course and is detrimental weight to women's quality of life, sexual function, and general health. IC/BPS affects nearly 1.2 million women in the United States and although there are currently six lines of treatment, they lack high level evidence and sufficient efficacy. New therapies are in high demand. As the cannabis industry gains popularity in medicine, research has revealed prevalent expression of cannabinoid receptors in bladder detrusor muscle and urothelium suggesting a novel drug target for IC/BPS. This study seeks to exploit this target by conducting a double-masked, placebo-controlled randomized trial evaluating the effects of vaginal hemp cannabidiol (CBD) suppositories on lower urinary tract symptoms (LUTS), pain severity, and sexual function. Women with diagnosed IC/BPS will be randomized to treatment with a placebo vaginal suppository or a hemp CBD vaginal suppository. We will monitor changes in their LUTS, pain, and sexual function using validated questionnaires. Our goal is to evaluate whether CBD is an effective, low-risk and less invasive treatment option for IC/BPS. Attainment of this goal would demonstrate a potential novel use for CBD in our Urogynecology patient population.

ELIGIBILITY:
Inclusion Criteria:

* Female Subjects ≥ 18 years of age
* Interstitial cystitis (IC) diagnosis
* English speaking/reading
* Prior treatment with one known treatment for IC: behavioral modifications, pelvic floor physical therapy, medications (amitriptyline, cimetidine, pentosane polysulfate sodium, or hydroxyzine), bladder instillations, bladder hydrodistention, cystoscopic fulguration or injection of Hunner's lesions, intradetrusor injection of botulinum toxin, or sacral neuromodulation
* Females of childbearing potential must use contraception throughout the study period (hormonal contraception, diaphragm, cervical cap, vaginal sponge, condoms, vasectomy, long acting reversible contraception)
* Females of non-child bearing potential must be post-menopausal defined as: > 51yo with no menses within the past 12mo or history of hysterectomy or history of bilateral oophorectomy or bilateral tubal ligation

Exclusion Criteria:

* THC or cannabidiol use within 1 month prior to enrollment per patient report
* Positive urine marijuana drug test on day of study enrollment
* Plan to use concomitant THC or cannabidiol of any form during the 6 week study period
* Inability to speak/understand English
* Pregnant or planning on becoming pregnant
* Unable to be contacted for follow up by telephone
* Cocoa butter allergy
* AST or ALT greater than 3 times the upper limit of normal at time of enrollment
* Females of childbearing potential with a positive urine pregnancy test at screening/prior to administration of Day 1 of treatment
* Subjects taking prescription or non-prescription medication which are substrates of CYP3A4, CYP2C19, CYP2C8, CYP2C9, CYP2C19, CYP1A2 and CYP2B6 within 14 days of the study procedure

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Urinary Pain Severity Scores | 6 weeks
  Compare the efficacy of vaginal CBD suppositories versus vaginal placebo suppositories on pain severity symptoms in IC/BPS patients, as measured by composite pain severity sub-scores of the Genitourinary Pain Index (GUPI) & Interstitial Cystitis Symptom Index (ICSI). The score ranges from 0-27 composite score with higher scores being consistent with more symptomatic disease.

SECONDARY OUTCOMES:
Urinary Symptom Severity Scores | 6 weeks
  Compare the efficacy of vaginal CBD suppositories versus vaginal placebo suppositories on lower urinary tract symptoms as measured by the composite urinary severity sub-scores of the Genitourinary Pain Index (GUPI) & Interstitial Cystitis Symptom Index (ICSI). The score ranges from 0-25 composite score with higher scores being consistent with more symptomatic disease.
Marijuana Urine Drug Test | 6 weeks
  Evaluate the effect of routine use of vaginal CBD suppositories on a standard over-the-counter marijuana urine drug test

CONTACTS AND LOCATIONS:
Overall Officials: Gena Dunivan, M.D., Principal Investigator — University of New Mexico Department of Urogynecology
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No